CLINICAL TRIAL: NCT00732979
Title: IVC CLAMP: Infrahepatic Inferior Vena Cava Clamping During Hepatectomy - A Randomized Controlled Trial
Brief Title: Infrahepatic Inferior Vena Cava Clamping During Hepatectomy
Acronym: IVC CLAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Nuh Rahbari, MD, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NNR-01
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Hemorrhage
Keywords: Elective; hepatic; resection; due to any; reason.
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Infrahepatic inferior vena cava clamping The inferior vena cava is circumferentially dissected below the liver and clamped with a vascular clamp. Patients in this study group will receive intravenous volume for maintenance of fluid hemostasis according to local standards.
  Interventions: Procedure: Infrahepatic inferior vena cava clamping
- B (Active Comparator): Patients in this study group undergo hepatic resection following current standards of the Departments of Surgery and Anesthesiology, University of Heidelberg. Current practice consists of no type of vascular control in combination with CVP reduction below < 5mmHg. CVP reduction is mainly attained using restricted intravenous fluid administration.
  Interventions: Procedure: No infrahepatic inferior vena cava clamping

INTERVENTIONS:
Procedure: Infrahepatic inferior vena cava clamping — The inferior vena cava is circumferentially dissected below the liver and clamped with a vascular clamp. Patients in this study group will receive intravenous volume for maintenance of fluid hemostasis according to local standards.
  Arms: A
Procedure: No infrahepatic inferior vena cava clamping — Patients in this study group undergo hepatic resection following current standards of the Departments of Surgery and Anesthesiology, University of Heidelberg. Current practice consists of no type of vascular control in combination with CVP reduction below < 5mmHg. CVP reduction is mainly attained using restricted intravenous fluid administration.
  Arms: B

SUMMARY:
Intraoperative blood loss is a major concern during hepatic resection, as it has been shown to adversely affect patients' perioperative outcome. Reduction of central venous pressure during parenchymal transection has been shown to effectively lower liver hemorrhage. While CVP reduction is mainly achieved via fluid restriction and diuretics, dehydration may impair organ function. Moreover, it may lead to hemodynamic instability, particularly in case of severe bleeding. For this reason the technique of infrahepatic inferior vena cava clamping has been suggested which is able to lower CVP without the need for fluid restriction.

In the present study the two strategies to reduce CVP and by this intraoperative bleeding, namely fluid restriction and inferior vena cava clamping are compared with intraoperative blood loss as primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years
* Scheduled for elective hepatic resection due to any reason
* American Society of Anesthesiologists (ASA) score I to III
* Written informed consent

Exclusion Criteria:

* Medical conditions exposing patient at increased risk for not tolerating liver resection:
* Cirrhosis (Child-Pugh B and C)
* (Hereditary) coagulopathy
* Medical conditions exposing patient at increased risk for not tolerating this trial's study interventions:
* Severe heart disease (e.g. severe CAD requiring intervention, NYHA IV)
* Pulmonary hypertension
* Renal insufficiency (serum creatinin >2mg/dl or >177µmol/l; conversion factor 88.4 or requiring dialysis)
* Severe hypernatremia (serum sodium >155mmol/l)
* Severe hyperchloremia
* For female subjects: pregnancy and lactation
* Impaired mental state or language problems
* Participation in other clinical trials or observation period of competing trials interfering with the endpoints of this trial
* Former participation in the clinical trial
* Expected lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2008-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | End of operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General, Visceral and Transplantation Surgery, University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Rahbari NN, Koch M, Zimmermann JB, Elbers H, Bruckner T, Contin P, Reissfelder C, Schmidt T, Weigand MA, Martin E, Buchler MW, Weitz J. Infrahepatic inferior vena cava clamping for reduction of central venous pressure and blood loss during hepatic resection: a randomized controlled trial. Ann Surg. 2011 Jun;253(6):1102-10. doi: 10.1097/SLA.0b013e318214bee5. PMID 21412143
- [Derived] Rahbari NN, Zimmermann JB, Koch M, Bruckner T, Schmidt T, Elbers H, Reissfelder C, Weigand MA, Buchler MW, Weitz J. IVC CLAMP: infrahepatic inferior vena cava clamping during hepatectomy--a randomised controlled trial in an interdisciplinary setting. Trials. 2009 Oct 13;10:94. doi: 10.1186/1745-6215-10-94. PMID 19825186